CLINICAL TRIAL: NCT05174897
Title: The Effect of Emotional Freedom Technique Used in Intravenous Catheter Applications in Pediatric Emergency on Fear and Pain
Brief Title: The Effect of Emotional Freedom Technique on Fear and Pain in Intravenous Catheter Applications in Pediatric Emergency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Müge SEVAL (Other)
Responsible Party: Sponsor-Investigator, Müge SEVAL, Doctoral Lecturer, Zonguldak Bulent Ecevit University
Organization: Zonguldak Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/20-9
Record Dates: First submitted 2021-11-18; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Pain; Fear
Keywords: Emotional Liberation Technique; intravenous catheter; child emergency
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled study to examine the effect of the emotional freedom technique used in intravenous catheter applications in the pediatric emergency on fear and pain in children aged 10-14 years. The entire sample was numbered from 1 to 70, and odd numbers were assigned to the control group and even numbers to the intervention group. Randomization was performed by an independent nurse other than the researcher.
Who Masked: Outcomes Assessor
Masking Description: The aim of this study is to evaluate the effect of emotional liberation technique (EFT) in reducing fear and pain during intravenous catheterization in children aged 10-14 years who applied to the emergency department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The child for whom an intravenous catheter will be applied will be placed on a stretcher and pain and fear will be evaluated before the procedure. Afterwards, an intravenous catheter will be applied. Pain and fear scores will be evaluated during and after the procedure.
- Experimental group (Experimental): The child to whom an intravenous catheter will be applied is placed on a stretcher. After evaluating the pain and fear score before the procedure, emotional liberation technique (EFT) is performed for 10 minutes. followed by an intravenous catheter. Pain and fear scores are evaluated during and after the procedure.
  Interventions: Behavioral: emotional liberation technique

INTERVENTIONS:
Behavioral: emotional liberation technique — experimental group; The child, to whom an intravenous catheter will be applied, is placed on a stretcher. pain ve score fear will be evaluated before the procedure. Then, the emotional liberation technique (EFT) will be applied for 10 minutes and an intravenous catheter will be applied to evaluate the pain and fear scores during and after the procedure.
  Arms: Experimental group

SUMMARY:
This study was planned to determine the effect of emotional liberation technique (EFT) in reducing fear and pain in intravenous catheter applications in children aged 10-14 years admitted to the pediatric emergency department.

DETAILED DESCRIPTION:
Emotional Freedom Technique is an easy-to-apply therapy method, which is one of the energy psychotherapy methods. The basic principle of the technique is that every limiting thought, disturbing emotion and memory that the individual has is related to the disruption of the electrical flow in his body and creating congestion.

When children apply to the hospital due to illness, they feel anxiety, fear and are exposed to unpleasant procedures that disturb them. Illness and hospitalization cause trauma for children of all age groups. However, there are negative effects on the development of children. Experiencing negative physical events, undergoing surgery and separation of children from their families is a difficult process for them. Children who experience negative emotions during this difficult process also worry about physical limitations. In this case, unlike other friends, they may feel inadequate and blocked. Children experience more uncertain feelings about all procedures to be performed in the hospital than adults. The fact that children have to be in the hospital causes them to experience physiological, emotional and behavioral problems. In these cases, it is important to reduce the negative effects of hospital admissions on children.

Pediatric pain itself is a problem for a child, their parents, and medical staff in a pediatric emergency room. Studies have shown that up to 80% of emergency room patients undergo painful diagnostic procedures such as vein puncture, intravenous insertion and removal, tape removal, and urine sampling. Painful procedures are often unexpected. It therefore intensifies the stress and anxiety associated with the hospital, leading to unpleasant experiences and bad memories associated with medical settings that can adversely affect procedure results. It can also affect future visits and increase the patient's fears. The simple thought of visiting hospital settings can also be distressing for a child. A crowded emergency room environment can be a source of fear and anxiety for children. Children's age and gender, development and communication level, different personalities and temperaments, individual clinical situation and personal response to a painful stimulus should also be addressed. However, studies in the literature on reducing the anxiety and fears of children in the pediatric emergency service were also found to be insufficient.

It is the pain that children are most exposed to in hospitals and during the interventional procedures they do not want. According to the definition of the International Pain Research Organization, pain is; They are unpleasant, sensory and emotional states that are affected by the past experiences of individuals resulting from actual or potential tissue damege. Each child perceives and expresses pain differently. Pain control in children begins with the assessment of pain. Afterwards; Relief of the child's pain and the ability to cope with pain increase the quality of life is provided. Although it is preferred because we all know about the control of pain and the effect of pharmacological methods is seen quickly with its easy applicability, excessive and unconscious use affects physiological functions negatively. Today, although its use has increased compared to the past, non-pharmacological methods that have not reached a sufficient level can be applied easily without harming the body. It can also be applied in pain management by increasing the release of endorphins, the body's natural morphine. There are many non-pharmacological methods that can be applied to us. One of them is acupressure applications. With the acupressure application, gentle strokes are made on the acupuncture points in the body. With these touches, the nociception process begins and the impulses stimulate the serotoninergic and enkephalinergic agents to activate the analgesic system.

An EFT tour is carried out by making light strokes on the transit points of the 14 main meridians in the body. The basic application of EFT is respectively; It starts with the determination of the subjective discomfort level Subjective Units of Disturbance/ SUD. Here on a scale from -10 to +10; -10 of the greatest pain, fear, stress and sadness imaginable; +10 allows us to evaluate the scaling that includes the highest levels of joy, happiness, and well-being. Next, the preparation or setup sentence is formed and repeated by rubbing the space between the chest and shoulder. The sentences are repeated and the acupuncture points are hit in order. After the EFT tour, it is evaluated whether there is a difference in the level of discomfort of the individual with the SUD scale. When measured against the standards of the American Psychological Association's Chapter 12 Task Force on Empirically Validated Therapies, EFT has been found to be an evidence-based practice for anxiety, depression, phobias, and post-traumatic stress disorder.

When the literature studies are examined; Positive results of EFT were obtained and no side effects were observed. Emotional liberation techniques are used in children with test anxiety, fear, bedwetting, nightmares, sleep disorders, stress, school problems, learning difficulties and problems related to self-esteem. A study was conducted on the severity of venipuncture pain in hospitalized children aged 6-12 in Iran, comparing acupressure and topical anesthesia applications to Yintang and Laogong points. As a result of the study, it was seen that acupressure was as effective as topical anesthetic cream in relieving venipuncture pain in children. At the same time, the study suggests the use of acupressure practice in nurses' pediatric clinical. In another study example; Acupressure was applied 10 minutes before the venipuncture application and it was found to be effective in reducing the pain experienced by children. In another study example, the effect of acupressure on pain after tonsillectomy in adolescents. evaluated. In a study conducted with 144 children aged 5-12 years, it was observed that acupressure had a positive effect on reducing pain after tonsillectomy surgery.

It has also proven to be a noninvasive, safe and effective method. The use of studies in clinics is recommended and their dissemination should be ensured.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 10-14
* The child is awake/cooperative
* No life-threatening condition/No medical contraindications
* Absence of physical/mental/cognitive development problems Having one of the diagnoses of fever, bronchitis/asthma, nausea-vomiting, abdominal pain, allergy
* The child's willingness and declaring it in writing
* Children of families who signed the informed consent form by accepting to participate in the study will be included in the study.

Exclusion Criteria:

* not be between the ages of 10-14
* The child is not alert/cooperative
* There is a life-threatening condition/There is a medical contraindication
* Having a physical/mental/cognitive development problem Not having one of the diagnoses of fever, bronchitis/asthma, nausea-vomiting, abdominal pain, allergy
* The child does not want to participate in the study
* families' refusal to work

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Pen Pain Scale | 0-2 years
  It will be used to measure the pain scores of children in the experimental and control groups before, during and after the procedure. The pencil used as a scale is a handmade pencil whose raw material is wood and measures 17 cm in length, 5 cm in circumference and 1.59 cm in diameter. In the middle of the pen, a monthly 5 cm long, parallel to its neck, is formed and drawn in orange around it to be decisive. A 5 cm measurement line was drawn by hand in the middle of the recess and is numbered from 0 to 5. While the value near the tip of the pen indicates 0 and the value near the base indicates 5, the value 0 means no pain and 5 means unbearable pain.
Medical Procedures Fear Scale | 0-2 years
  Medical Procedures Fear Scale It will be used to calculate the fear scores of the children in the experimental and control groups before, during and after the procedure. The scale items were prepared in the form of a structured Likert-type 3-point timed option, and the child was required to choose one of the statements 'I am not afraid at all', 'I am somewhat afraid', 'I am very afraid' for each item. Scores range from 29 to 87, and those with low scores constitute the group that is least afraid of medical procedures.
Subjective Experience Scale(SUE) | 0-2 years
  As the subjective scoring of the experience, it will be applied to the children in the experimental group before and after the procedure. An SUE assessment is done before the EFT round begins. After the EFT round is complete, the SUE scale is repeated to see how much the situation has changed. on a scale from -10 to +10; -10 indicates the greatest imaginable level of pain, frustration, fear, stress, sadness, or discomfort. +10; It includes the highest levels of joy, happiness, or feeling great.
Heart rate | 0-2 years
  The heart rate of the children was recorded by measuring with a pulse oximeter placed on the right or left finger of each child. Heart rate was recorded before, during and after the procedure.
oxygen saturation | 0-2 years
  The oxygen saturation value of the children was measured with a pulse oximeter placed on the right or left finger of each child and recorded. Oxygen value was recorded before, during and after the procedure.
respiratory rate | 0-2 years
  The respiratory rate of the children was evaluated by the researcher within one minute. Respiratory values were recorded before, during and after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin KARAMAN, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No